CLINICAL TRIAL: NCT01277679
Title: An Evaluation of MRI Measures of Lung Water Increases With Postural Changes in Healthy Subjects and in Patients With Cardiac Failure: A Methods Validation Study for Evaluation of Novel Treatments Limiting Pulmonary Oedema in Cardiac Failure
Brief Title: Evaluation of MRI Measures of Lung Water With Posture Changes in Healthy Volunteers and in Patients With Cardiac Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 114747
Record Dates: First submitted 2010-11-18; First posted 2011-01-17 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure, Congestive
Keywords: lung water measures; pulmonary edema; MRI; heart failure
MeSH Terms: conditions — Heart Failure; Pulmonary Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteer (Other): Healthy Volunteer cohort
  Interventions: Procedure: MRI
- Heart Failure (Other): Heart Failure cohort
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI of lungs to measure lung water content before and after passive leg raising (PLR)

SUMMARY:
The aim of this study is to establish a model for the evaluation of drug targets using postural measures to induce changes in lung water concentration as assessed by MRI. A reduction in the magnitude and rate of water transudation with postural changes in patients with congestive heart failure (CHF) could provide a model for the evaluation of various classes of molecules for target validation and for dose selection.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure Patients:
* Established diagnosis of mild to moderate heart failure of any aetiology with symptoms defined as corresponding to the New York Heart Association (NYHA) class I, II or III
* Able in the opinion of the patient and investigator to be supine for 1 hour and to experience passive leg raising (PLR) whilst in the MRI scanner
* Male or female over 18 years of age at the time of signing the informed consent
* Negative urine or serum pregnancy test
* Capable of giving written informed consent
* Registered with a UK general practitioner.
* Participants must read (in English) at a level sufficient to adequately complete study related questionnaires
* Able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* Healthy Volunteers:
* Healthy as determined by a responsible physician
* Male or female over 18 years of age at the time of signing the informed consent
* Capable of giving written informed consent
* Negative urine or serum pregnancy test
* Registered with a UK general practitioner
* Participants must read (in English) at a level sufficient to adequately complete study related questionnaires
* Able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Exclusion Criteria:

* Heart Failure Patients
* History of primary pulmonary disease requiring current medication or other therapy.
* Orthopnoea of sufficient severity to preclude supine scanning.
* Hip or leg pathology of sufficient severity to prevent extension of both legs to 45 degrees.
* Unstable heart failure, defined as change in NYHA status, change in heart failure therapy regimen or hospitalization for acute decompensation of heart failure within preceding 6 weeks.
* Unstable angina within the past 3 months
* Current smoker, defined as having smoked in the preceding 1 year
* Uncontrolled hypertension (resting systolic BP > 160 mmHg or resting diastolic BP > 100mmHg)
* Resting hypoxia (SaO2 <93%).
* Contraindication to MRI scanning
* Pregnant females
* Positive drugs of abuse or alcohol screen.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Healthy Volunteers
* History of primary pulmonary disease requiring current medication or other therapy
* Current smoker, defined as having smoked in the preceding 1 year
* Hip or leg pathology of sufficient severity to prevent extension of both legs to 45 degrees
* Contraindication to MRI scanning
* Pregnant females
* Positive drugs of abuse or alcohol screen
* Unwillingness or inability to follow the procedures outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Lung water distribution as measured by MRI | Visit 1 and Visit 2 will be approximately 1 week apart
  MRI test
Lung water concentration as measured by MRI | Visit 1 and Visit 2 will be approximately 1 week apart
  MRI test

SECONDARY OUTCOMES:
Between patient variability in lung water concentration as measured by MRI at 2 independent visits | Visit 1 and Visit 2 will be approximately 1 week apart
  MRI test
Within patient variability in lung water concentration as measured by MRI at 2 independent visits | Visit 1 and Visit 2 will be approximately 1 week apart
  MRI test

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom